CLINICAL TRIAL: NCT02912728
Title: Strategies to Enhance New CGM Use in Early Childhood: A Randomized Clinical Trial to Assess the Efficacy and Safety of Continuous Glucose Monitoring in Youth < 8 With Type 1 Diabetes
Brief Title: Strategies to Enhance New CGM Use in Early Childhood (SENCE)
Acronym: SENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: The Leona M. and Harry B. Helmsley Charitable Trust (Other); Indiana University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: T1DX SENCE
Record Dates: First submitted 2016-09-20; First posted 2016-09-23 (Estimated); Last update posted 2020-10-05 (Actual); Status verified 2020-10

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- CGM + Family Behavioral Intervention (Active Comparator): CGM training for CGM groups using a standard curriculum will take place at the 1, 3 and 6 week visits in addition to the training at baseline. The family behavioral intervention will be delivered by a study coordinator (separate coordinator from the CGM instruction) at the 1, 3, 6, 13 and 19 week visits and is expected to take approximately 30 minutes.
  Interventions: Behavioral: CGM + Family Behavioral Intervention
- Standard CGM (Active Comparator): Each participant will be asked to use a CGM sensor on a daily basis, inserting a new sensor as needed with a maximum of 7 days of wear per sensor.
  A home BGM will be used for calibration of the CGM sensor. Additional BGM glucose measurements may be performed by the participant at any time, particularly prior to making a real-time management decision based on the CGM glucose reading.
  Participants will be instructed to use the CGM as per the FDA labeling.
  Interventions: Device: Standard CGM
- BGM - usual care control group (No Intervention): A BGM will be used for a finger stick blood glucose check with a recommendation of at least 4 times a day. BGM data will be downloaded and reviewed with the participant at each visit.

INTERVENTIONS:
Behavioral: CGM + Family Behavioral Intervention — use of CGM combined with a CGM focused family behavioral intervention and to assess CGM adherence
  Other Names: FBI
  Arms: CGM + Family Behavioral Intervention
Device: Standard CGM — use of CGM alone to assess CGM adherence
  Arms: Standard CGM

SUMMARY:
The primary objective of this study is to compare the efficacy and safety of CGM alone and CGM combined with a family behavioral intervention with a control group using home blood glucose monitoring (BGM) alone.

DETAILED DESCRIPTION:
Although prior studies have not demonstrated that continuous glucose monitoring (CGM) use results in improved glycemic control in children <8 years of age, many of the barriers to CGM efficacy in this age group may have been due to problems in the wearability and accuracy of prior generation devices, as well as to the setting of glycemic targets aimed primarily at preventing hypoglycemia at all costs. There may also be behavioral barriers to consistent and effective CGM use in this age range. The goal of this study is to assess the impact of CGM alone and CGM combined with a family behavioral intervention focused on supporting CGM use on glycemic control in very young children with T1D compared with usual care without CGM.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of insulin dependent presumed autoimmune type 1 diabetes by the investigator
2. Age 2-<8 years at consent
3. Diabetes duration ≥ 6 months
4. Total daily insulin ≥ 0.3 units per kg per day
5. HbA1c 7.0% to <10.0% (Point of care device or local lab measured within 30 days of screening visit used to assess eligibility)
6. No use of unblinded personal CGM, outside of a research study, as part of real-time diabetes management in the last 30 days
7. Insulin regimen involves either use of a consistent insulin regimen with an insulin pump in the last 3 months or at least 3 multiple daily injections of basal and bolus (meal time) analogue insulin in the last 3 months (e.g. no change from injections to pump or vice versa in the last 3 months), with no plans to switch the modality of insulin administration during the next 6 months (e.g., injection user switching to a pump, pump user switching to injections).
8. Perform at least 3 blood glucose meter checks per day from self-report at screening and meter download during blinded CGM run in
9. Not currently using and no plans to begin non-insulin medication for blood glucose lowering during the course of the study
10. Parent or guardian comprehend written and spoken English (This requirement is due to the fact that the questionnaires to be used as outcome measures do not have validated versions in other languages, and interventions will be delivered in English only for the RCT to ensure standardization/fidelity checks across sites).
11. Parent understands the study protocol and agrees to it
12. No expectation that participant/parent will be moving out of the area of the clinical center during the next 12 months, unless the move will be to an area served by another study center.

Exclusion Criteria:

1. Use of unblinded personal CGM, outside of a research study, as part of real-time diabetes management in the last 30 days
2. Unable to use CGM device for minimum number of hours during blinded run-in period or skin reaction from adhesive that would preclude participation in the randomized trial
3. The presence of a significant medical disorder or use of a medication such as oral/inhaled glucocorticoids that in the judgment of the investigator will affect the wearing of the sensors or the completion of any aspect of the protocol.
4. More than 1 episode of SH or DKA in the past 6 months (not including DKA at time of dx).
5. The presence of any of the following diseases:

   * Asthma if treated with systemic or daily inhaled corticosteroids in the last 6 months (Intermittent treatment with inhaled corticosteroids does not exclude subjects from enrollment)
   * Cystic fibrosis (Adequately treated thyroid disease and celiac disease do not exclude subjects from enrollment)
6. Inpatient psychiatric treatment in the past 6 months for either child participant or the primary care giver
7. Need for use of acetaminophen or acetaminophen-containing products on a regular basis during the 6 months of the trial
8. Participation of parent or child in a diabetes related intervention study in past 6 weeks.
9. Any medical, psychological or social situation where per investigator discretion it may be difficult for family or child to participate fully in the intervention
10. Another member of the same household is participating in this study.

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 143 (Actual)
Dates: Start 2017-01-30 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Time in glucose range 70-180 | Up to 26 weeks
  The primary outcome will be three 2 group comparisons of the change from baseline in the percentage of sensor values in the target range (70-180 mg/dL), in an ANCOVA model adjusted for the baseline value and factors used to stratify randomization with clinical site as a random effect. Seven days of sensor glucose values during the week prior to the 6, 13, 19 and 26 week clinic visits will be used in analysis for the CGM groups to match up with the blinded CGM placed at each visit in the control group. The CGM data will be pooled across each visit where CGM data are collected during follow up for the primary analysis.

SECONDARY OUTCOMES:
HbA1c at 6-months | 6 Months
  A secondary outcome is to compare HbA1c at 6-months, adjusted for baseline.
% HbA1c <7.0% | 6 Months
% HbA1c <7.5% | 6 Months
% with relative reduction in HbA1c >=10% | 6 Months
% with absolute reduction in HbA1c >=0.5% | 6 Months
% with absolute reduction in HbA1c >=1% | 6 Months
% with absolute reduction in HbA1c >=1% or HbA1c <7.0% | 6 Months
Mean glucose | 6 Months
Glucose variability measured by coefficient of variation | 6 Months
% time >180 mg/dl | 6 Months
% time >250 mg/dl | 6 Months
% time >300 mg/dl | 6 Months
Area under the curve 180 mg/dl | 6 Months
High blood glucose index (HBGI) | 6 Months
% time <54 mg/dl | 6 Months
% time <60 mg/dl | 6 Months
% time <70 mg/dl | 6 Months
Area over the curve 70 mg/dl | 6 Months
Low blood glucose index (LBGI) | 6 Months
Hypoglycemic events (using <54 mg/dl) | 6 Months
WHO-5 Well Being Index | 6 Months
  Survey containing 5 questions with possible responses 0-5. The raw score is calculated by summing the responses. The raw score ranges from 0-25. A percentage score ranging from 0 to 100 is obtained by multiplying the raw score by 4. A percentage score of 0 represents worst possible, whereas a score of 100 represents best possible quality of life.
Hypoglycemia Fear Survey Total Score | 6 Months
  Survey containing 26 questions with possible responses 0-4. Total score is calculated by taking the mean of the non-missing responses and multiplying by 25 to put on the scale 0-100. A higher score indicates more fear.
Hypoglycemia Fear Survey Worry Subscale | 6 Months
  Survey containing 26 questions with possible responses 0-4. Worry subscale score is calculated by taking the mean of the non-missing responses to questions 11-26 and multiplying by 25 to put on the scale 0-100. A higher score indicates more fear.
Diabetes Technology Questionnaire | 6 Months
  Survey containing 30 questions with possible responses 0-4. Total score is calculated by taking the mean of the non-missing responses and multiplying by 100 to put on the scale 0-100. A higher total score indicates less of a problem.
Problem Areas in Diabetes - Parent (PAID-PR) | 6 Months
  Survey containing 18 questions with possible responses 0-4. Total score is calculated by reverse scoring each item, then taking the mean of the non-missing responses. The score is then multiplied by 25 to put on the scale 0-100. A higher total score indicates more burden.
Diabetes Family Impact Survey | 6 Months
  Survey containing 15 questions with possible responses 0-3. Total score is calculated by taking the mean of the non-missing responses. Then multiply by 100 and divide by 3 to put on the scale 0-100. A higher total score indicates more negative impact.
Satisfaction Questionnaire | 6 Months
  Section 2 of the satisfaction questionnaire contains 8 questions for the CGM groups only with possible responses 0-4. Total score is calculated by taking the mean of the non-missing responses and multiplying by 25 to put on the scale 0-100. A higher total score indicates more satisfaction with the study.

CONTACTS AND LOCATIONS:
Overall Officials: Linda DiMeglio, MD, MPH, Principal Investigator — Indiana University School of Medicine
Locations (1):
- Indiana, Indianapolis, Indiana, United States

REFERENCES:
- [Background] Mauras N, Beck R, Xing D, Ruedy K, Buckingham B, Tansey M, White NH, Weinzimer SA, Tamborlane W, Kollman C; Diabetes Research in Children Network (DirecNet) Study Group. A randomized clinical trial to assess the efficacy and safety of real-time continuous glucose monitoring in the management of type 1 diabetes in young children aged 4 to <10 years. Diabetes Care. 2012 Feb;35(2):204-10. doi: 10.2337/dc11-1746. Epub 2011 Dec 30. PMID 22210571
- [Background] Sundberg F, Forsander G. Detection and treatment efficacy of hypoglycemic events in the everyday life of children younger than 7 yr. Pediatr Diabetes. 2014 Feb;15(1):34-40. doi: 10.1111/pedi.12057. Epub 2013 Jun 27. PMID 23809540
- [Background] Rovet JF, Ehrlich RM. The effect of hypoglycemic seizures on cognitive function in children with diabetes: a 7-year prospective study. J Pediatr. 1999 Apr;134(4):503-6. doi: 10.1016/s0022-3476(99)70211-8. PMID 10190928
- [Background] Rovet JF, Ehrlich RM, Hoppe M. Specific intellectual deficits in children with early onset diabetes mellitus. Child Dev. 1988 Feb;59(1):226-34. doi: 10.1111/j.1467-8624.1988.tb03211.x. PMID 3342715
- [Background] Ryan CM. Searching for the origin of brain dysfunction in diabetic children: going back to the beginning. Pediatr Diabetes. 2008 Dec;9(6):527-30. doi: 10.1111/j.1399-5448.2008.00481.x. No abstract available. PMID 19067890
- [Background] Barnea-Goraly N, Raman M, Mazaika P, Marzelli M, Hershey T, Weinzimer SA, Aye T, Buckingham B, Mauras N, White NH, Fox LA, Tansey M, Beck RW, Ruedy KJ, Kollman C, Cheng P, Reiss AL; Diabetes Research in Children Network (DirecNet). Alterations in white matter structure in young children with type 1 diabetes. Diabetes Care. 2014 Feb;37(2):332-40. doi: 10.2337/dc13-1388. Epub 2013 Dec 6. PMID 24319123
- [Background] Marzelli MJ, Mazaika PK, Barnea-Goraly N, Hershey T, Tsalikian E, Tamborlane W, Mauras N, White NH, Buckingham B, Beck RW, Ruedy KJ, Kollman C, Cheng P, Reiss AL; Diabetes Research in Children Network (DirecNet). Neuroanatomical correlates of dysglycemia in young children with type 1 diabetes. Diabetes. 2014 Jan;63(1):343-53. doi: 10.2337/db13-0179. Epub 2013 Oct 29. PMID 24170697
- [Background] Wood JR, Miller KM, Maahs DM, Beck RW, DiMeglio LA, Libman IM, Quinn M, Tamborlane WV, Woerner SE; T1D Exchange Clinic Network. Most youth with type 1 diabetes in the T1D Exchange Clinic Registry do not meet American Diabetes Association or International Society for Pediatric and Adolescent Diabetes clinical guidelines. Diabetes Care. 2013 Jul;36(7):2035-7. doi: 10.2337/dc12-1959. Epub 2013 Jan 22. PMID 23340893
- [Background] Tsalikian E, Fox L, Weinzimer S, Buckingham B, White NH, Beck R, Kollman C, Xing D, Ruedy K; Diabetes Research in Children Network Study Group. Feasibility of prolonged continuous glucose monitoring in toddlers with type 1 diabetes. Pediatr Diabetes. 2012 Jun;13(4):301-7. doi: 10.1111/j.1399-5448.2011.00837.x. Epub 2011 Dec 13. PMID 22151826
- [Background] Topp CW, Ostergaard SD, Sondergaard S, Bech P. The WHO-5 Well-Being Index: a systematic review of the literature. Psychother Psychosom. 2015;84(3):167-76. doi: 10.1159/000376585. Epub 2015 Mar 28. PMID 25831962
- [Background] Markowitz JT, Volkening LK, Butler DA, Antisdel-Lomaglio J, Anderson BJ, Laffel LM. Re-examining a measure of diabetes-related burden in parents of young people with Type 1 diabetes: the Problem Areas in Diabetes Survey - Parent Revised version (PAID-PR). Diabet Med. 2012 Apr;29(4):526-30. doi: 10.1111/j.1464-5491.2011.03434.x. PMID 21883443
- [Background] Katz ML, Volkening LK, Dougher CE, Laffel LM. Validation of the Diabetes Family Impact Scale: a new measure of diabetes-specific family impact. Diabet Med. 2015 Sep;32(9):1227-31. doi: 10.1111/dme.12689. Epub 2015 Feb 5. PMID 25655562
- [Background] Cox DJ, Irvine A, Gonder-Frederick L, Nowacek G, Butterfield J. Fear of hypoglycemia: quantification, validation, and utilization. Diabetes Care. 1987 Sep-Oct;10(5):617-21. doi: 10.2337/diacare.10.5.617. PMID 3677982
- [Background] Wysocki T, Reeves G, Kummer M, Ross J, Yu M. Psychometric validations of the Diabetes Technology Questionnaire; Diabetes. 2015;64(Suppl1): A633.
- [Derived] Strategies to Enhance New CGM Use in Early Childhood (SENCE) Study Group. A Randomized Clinical Trial Assessing Continuous Glucose Monitoring (CGM) Use With Standardized Education With or Without a Family Behavioral Intervention Compared With Fingerstick Blood Glucose Monitoring in Very Young Children With Type 1 Diabetes. Diabetes Care. 2021 Feb;44(2):464-472. doi: 10.2337/dc20-1060. Epub 2020 Dec 17. PMID 33334807
- [Derived] DiMeglio LA, Kanapka LG, DeSalvo DJ, Anderson BJ, Harrington KR, Hilliard ME, Laffel LM, Tamborlane WV, Van Name MA, Wadwa RP, Willi SM, Woerner S, Wong JC, Miller KM; SENCE Study Group. Time spent outside of target glucose range for young children with type 1 diabetes: a continuous glucose monitor study. Diabet Med. 2020 Aug;37(8):1308-1315. doi: 10.1111/dme.14276. Epub 2020 Mar 17. PMID 32096282